CLINICAL TRIAL: NCT04715841
Title: Gait Analysis in Females Suffering From Patellofemoral Pain Syndrome (PFPS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, walaa eldesoukey heneidy, lecturer of physical therapy, Delta University for Science and Technology
Other Study IDs: PFPS
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: Group A (Study group ) : 25 adolescent females suffering patellofemoral pain syndrome were recruited from the outpatient clinic of the faculty of physical therapy delta university in addition to the medical diagnosis was confirmed by consultant orthopedist using clinical and radiographic investigations .
  Interventions: Other: gait assessment
- group B: Group B (Control Group):25 adolescent females with healthy knee joints with no clinical and radiographic evidence of patellofemoral pain syndrome , were recruited from the students of the faculty of physical therapy delta university .
  Interventions: Other: gait assessment

INTERVENTIONS:
Other: gait assessment — gait assessment were done using 3DMA system

SUMMARY:
The purpose of the study was to evaluate the spatial and temporal variables during walking cycle in adolescent females suffering from patellofemoral pain syndrome (PFPS) versus healthy adolescent females .

ELIGIBILITY:
Inclusion Criteria:

* peripatellar or retropatellar knee pain worsen with upstairs and walking

Exclusion Criteria:

* previous knee or patella surgeries

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: 50 female with patellofemoral pain syndrome aged from 18 to 35 years old free from any musculoskeletal problems in lower limb
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
step length | 3 months
  measured during gait cycle in adolescent females suffering patellofemoral pain syndrome (PFPS) versus healthy adolescent females was done in motion analysis lab in Delta University for Science & Technology which equipped with walkway and six infrared cameras operating at 60 HZ frequency.
stride length | 3 months
  measured during gait cycle in adolescent females suffering patellofemoral pain syndrome (PFPS) versus healthy adolescent females was done in motion analysis lab in Delta University for Science & Technology which equipped with walkway and six infrared cameras operating at 60 HZ frequency.
speed | 3 months
  measured during gait cycle in adolescent females suffering patellofemoral pain syndrome (PFPS) versus healthy adolescent females was done in motion analysis lab in Delta University for Science & Technology which equipped with walkway and six infrared cameras operating at 60 HZ frequency.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Delta University for Science and Technology, Gamasa, Dakahelia
  - Delta University For Science and Technology, Gamasa

IPD SHARING:
Plan to Share IPD: No